CLINICAL TRIAL: NCT06876376
Title: Intraoperative Transvaginal and Endorectal Ultrasound for the Assessment of Bowel Deep Infiltrating Endometriosis
Brief Title: Intraoperative Ultrasound in Bowel Deep Endometriosis
Status: Recruiting | Type: Observational
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Sponsor
Other Study IDs: FSD-DIE-2024-18
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Deep Infiltrating Endometriosis With or Without Bowel Involvement
Keywords: Endometriosis; Intraoperative Ultrasound; Ultrasound; surgery; minimally invasive surgery
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- posterior compartment deep infiltrating endometriosis
  Interventions: Procedure: intraoperative ultrasound for the assessment of bowel deep infiltrating endometriosis

INTERVENTIONS:
Procedure: intraoperative ultrasound for the assessment of bowel deep infiltrating endometriosis — Women with posterior compartment deep infiltrating endometriosis with or without bowel involvement scheduled for surgical treatment at the Department of Obstetrics, Gynecology, and Reproductive Medicine of Dexeus University Hospital.

SUMMARY:
This study investigates the use of intraoperative transvaginal (IOTVUS) and/or endorectal ultrasound (IOERUS) in the surgical treatment of bowel deep infiltrating endometriosis (DIE).

DETAILED DESCRIPTION:
Bowel DIE is a severe form of endometriosis that often infiltrates the rectum and the sigmoid colon, requiring precise surgical techniques to achieve complete excision while minimizing unnecessary resections of healthy tissues and organs. Current preoperative imaging techniques, such as transvaginal ultrasound and magnetic resonance imaging, are often limited in their ability to assess lesion depth and extent in cases of severe pelvic anatomical distortion. Intraoperative ultrasound offers a real-time evaluation after rectal mobilization, allowing for a more accurate assessment of lesion location, depth, and bowel wall infiltration. The primary objectives are to evaluate the feasibility and accuracy of intraoperative ultrasound in detecting rectal and RSJ DIE nodules and to guide surgical decision-making. Secondary objectives include determining the impact of these techniques on surgical outcomes, postoperative pain management, and quality of life. The goal is to enhance surgical decision-making by accurately assessing lesion depth and location, potentially reducing unnecessary colorectal resections or avoiding inadvertent retention of endometrial nodules. Participants will complete health and pain questionnaires preoperatively and at 3, 6, and 12 months postoperatively, evaluating dysmenorrhea, dyspareunia, dyschezia, and quality of life using validated tools. The study will also document intraoperative findings, surgical decisions, complications, and postoperative outcomes. By combining IOTVUS and IOERUS with existing surgical approaches, this study seeks to establish these techniques as standard tools for improving surgical precision in bowel DIE cases. Results could provide valuable insights for tailoring interventions to patient-specific disease presentations, enhancing long-term management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative sonographic and/or MRI findings suggestive of bowel DIE (uterosacral ligaments, posterior vaginal wall, parametrium, retrocervical area, rectovaginal septum, rectum, and/or sigmoid colon).
* Scheduled for surgical treatment (laparoscopy or robot-assisted laparoscopy).
* Planned postoperative follow-up for at least 12 months.
* Written informed consent provided before surgery.

Exclusion Criteria:

* Planned surgery for diagnostic purposes only.
* Pregnancy at the time of enrollment.
* Poor understanding of Spanish or English.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with posterior compartment deep infiltrating endometriosis with or without bowel involvement scheduled for surgical treatment at the Department of Obstetrics, Gynecology, and Reproductive Medicine of Dexeus University Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intraoperative ultrasound | Day of surgery
  o The proportion of patients in whom intraoperative ultrasound techniques can successfully identify rectal or rectosigmoid junction deep infiltrating endometriosis nodules during surgery.
Accuracy of intraoperative ultrasound | Day of surgery
  o Agreement between intraoperative ultrasound findings and histopathological results regarding the depth of infiltration and size of bowel DIE nodules.

SECONDARY OUTCOMES:
Impact on Surgical Decision-Making | Day of surgery
  o Changes in surgical strategy (shaving, discoid excision, or segmental resection) based on intraoperative ultrasound findings.
Postoperative Pain and Function | at 3-months, 6-months and 12-months follow-up
  Improvement in pain symptoms and quality of life
Complication Rates | From day of surgery to 7 days later
  o Frequency of intraoperative or postoperative complications (ClassIntra and Clavien-Dindo ≥ III).

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Ginecología Obstetricia y Reproducción. Hospital Universitari Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giudice LC, Kao LC. Endometriosis. Lancet. 2004 Nov 13-19;364(9447):1789-99. doi: 10.1016/S0140-6736(04)17403-5. PMID 15541453
- [Background] Berkley KJ, Rapkin AJ, Papka RE. The pains of endometriosis. Science. 2005 Jun 10;308(5728):1587-9. doi: 10.1126/science.1111445. PMID 15947176
- [Background] de Ziegler D, Borghese B, Chapron C. Endometriosis and infertility: pathophysiology and management. Lancet. 2010 Aug 28;376(9742):730-8. doi: 10.1016/S0140-6736(10)60490-4. PMID 20801404
- [Background] Nnoaham KE, Hummelshoj L, Webster P, d'Hooghe T, de Cicco Nardone F, de Cicco Nardone C, Jenkinson C, Kennedy SH, Zondervan KT; World Endometriosis Research Foundation Global Study of Women's Health consortium. Impact of endometriosis on quality of life and work productivity: a multicenter study across ten countries. Fertil Steril. 2011 Aug;96(2):366-373.e8. doi: 10.1016/j.fertnstert.2011.05.090. Epub 2011 Jun 30. PMID 21718982
- [Background] Vercellini P, Vigano P, Somigliana E, Fedele L. Endometriosis: pathogenesis and treatment. Nat Rev Endocrinol. 2014 May;10(5):261-75. doi: 10.1038/nrendo.2013.255. Epub 2013 Dec 24. PMID 24366116
- [Background] Chapron C, Chopin N, Borghese B, Foulot H, Dousset B, Vacher-Lavenu MC, Vieira M, Hasan W, Bricou A. Deeply infiltrating endometriosis: pathogenetic implications of the anatomical distribution. Hum Reprod. 2006 Jul;21(7):1839-45. doi: 10.1093/humrep/del079. Epub 2006 Mar 16. PMID 16543256
- [Background] Scioscia M, Bruni F, Ceccaroni M, Steinkasserer M, Stepniewska A, Minelli L. Distribution of endometriotic lesions in endometriosis stage IV supports the menstrual reflux theory and requires specific preoperative assessment and therapy. Acta Obstet Gynecol Scand. 2011 Feb;90(2):136-9. doi: 10.1111/j.1600-0412.2010.01008.x. Epub 2010 Dec 2. PMID 21241258
- [Background] Donnez O, Roman H. Choosing the right surgical technique for deep endometriosis: shaving, disc excision, or bowel resection? Fertil Steril. 2017 Dec;108(6):931-942. doi: 10.1016/j.fertnstert.2017.09.006. PMID 29202966
- [Background] Abrao MS, Andres MP, Barbosa RN, Bassi MA, Kho RM. Optimizing Perioperative Outcomes with Selective Bowel Resection Following an Algorithm Based on Preoperative Imaging for Bowel Endometriosis. J Minim Invasive Gynecol. 2020 May-Jun;27(4):883-891. doi: 10.1016/j.jmig.2019.06.010. Epub 2019 Jun 22. PMID 31238150
- [Background] Puppo A, Olearo E, Gattolin A, Rimonda R, Novelli A, Ceccaroni M. Intraoperative Ultrasound for Bowel Deep Infiltrating Endometriosis: A Preliminary Report. J Ultrasound Med. 2021 Jul;40(7):1417-1425. doi: 10.1002/jum.15511. Epub 2020 Sep 29. PMID 32991006
- See also: Related Info — http://www.dexeus.com